ID: 2016-01

The Effect of Preoperative Ketamine on the Emergence Characteristics in Children Undergoing Entropion Surgery

NCT02916407

04-25-2019

We compared the emergence characteristics of sevoflurane versus desflurane with ketamine premedicated pediatric patients for ambulatory surgery. The primary outcome was compared the extubation time between sevoflurane versus desflurane anesthesia. The secondary outcome was compared the emergence characteristics (emergence agitation) between two groups.

Patients were randomly assigned into group S (sevoflurane) or group D (desflurane). After intravenous access in day-surgery unit, ketamine 1mg/kg was administered for separation from their parents, and then they were transferred to operating room with monitoring pulse oximetry. General anesthesia was maintained with sevoflurane in group S or desflurane in group D.

desflu

(MedCalor Su

a ± standhad dev

(interqua tile range,
as appropriate to compai

afficant. Data were analyzed using Medcalc 14.12.0 (MedCalc Software byba, Ostend, Belgium). Parametric variables were described as mean ± standard deviation (SD). Qualitative variables were described as number and as median (interquarule range). Student's t-test, Fisher's exact test, or Mann-Whitney U-test was used as appropriate to compare the two groups. P < 0.05 was